CLINICAL TRIAL: NCT01310244
Title: The Maximum Tolerated Dose and to Evaluate Safety and Efficacy of Belinostat (PXD-101) in Combination With Paclitaxel Plus Carboplatin in Chemotherapy-Naive Patients With Stage IV Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: MTD Study PXD-101 in Combination With Paclitaxel + Carboplatin in Chemotherapy-Naive Patients With Stage IV NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-1014-Bel
Record Dates: First submitted 2011-02-28; First posted 2011-03-08 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Stage IV Non-small Cell Lung Cancer
Keywords: Phase 1/2; MTD; stage IV; NSCLC; chemo-naive; Mixed-cell dose escalation; lung cancer; non-small-cell; phase I; Belinostat; Carboplatin; Paclitaxel; adenocarcinoma; PXD-101
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma | interventions — belinostat; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm, open label (Experimental): At the study entry each patient will receive a dose level assignment which will include a specific dose level and the dose of IV belinostat in mg/m2 to be administered during the study treatment.
  Belinostat will be infused over 30 minutes once daily on Days 1-5 of each 21-day cycle. On Day 3, the infusion of belinostat must be completed at least 1 hour prior to the start of the paclitaxel infusion. Dose of belinostat will be assigned at study entry. The same dose and level will remain throughout the entire study for each patient and no dose adjustment will be allowed, except due to toxicity.
  Interventions: Drug: Belinostat, Carboplatin, Paclitaxel

INTERVENTIONS:
Drug: Belinostat, Carboplatin, Paclitaxel — Up to 6 cycles of combination therapy of belinostat plus carboplatin (AUC 6) and paclitaxel 200 mg/m2. Initial dose of belinostat will be 1000mg/m2 for MTD dose escalation evaluation.
  Other Names: PXD-101

SUMMARY:
To define Phase 1/2 Maximum Tolerated Dose Study of Belinostat (PXD-101) in Combination with Paclitaxel plus Carboplatin in Chemotherapy-Naive Patients with Stage IV Non-Small-Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase 1/2, multi-center, open label single arm study. Patients meeting all inclusion and exclusion criteria will receive up to 6 cycles of combination therapy of belinostat plus carboplatin (AUC 6) and paclitaxel 200 mg/m2.

During phase I the Maximum Tolerated Dose (MTD) of belinostat in combination with carboplatin and paclitaxel will be determined in patients with Stage IV non-small cell lung cancer who have received no prior systemic chemotherapy. The dose escalation study will be conducted using traditional escalation rule of 3+3 design, during the first cycle of therapy. Belinostat will be assessed at a starting dose level of 1000 mg/m2 and multiple dose levels may be evaluated. Doses of belinostat, carboplatin and paclitaxel will remain constant throughout the study, unless dose modification is required by toxicity. Treatment is given on days 1-5 of every 21-day cycle. Routine safety evaluations will be conducted on days, 1, 8, and 15 of every cycle. Tumor measurement will be done after every 2 cycles of the treatment.

Additional 20 patients will be treated at the MTD defined dose during phase II expansion portion of the study.

All patients will receive up to 6 cycles of combination therapy and be followed until occurrence of unacceptable toxicity, disease progression, withdrawal of consent or death.

ELIGIBILITY:
Inclusion Criteria:

* A histologically or cytologically confirmed diagnosis of Stage IV (M1a or M1b) NSCLC. Patients with mixed non-small cell histologies are eligible
* No prior chemotherapy for the treatment of advanced NSCLC
* Prior adjuvant therapy for early stage lung cancer is allowed if completed ≥ 12 months prior to enrollment
* Age >= 18 years
* Adequate organ function
* Any treatment with investigational agent must have completed ≥ 4 weeks prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Negative pregnancy test for women of childbearing potential.
* Patients with brain metastases allowed if:

  * Directed local therapy was completed 2 weeks prior to enrollment;
  * There is no evidence of disease progression and;
  * Steroids are not required

Exclusion Criteria:

* Patients with mixed tumors of small cell features
* Known infection with HIV, hepatitis B or hepatitis C
* Baseline prolongation of QT/QTcF interval or required concomitant medication that may cause Torsade de Pointes
* Preexisting ≥Grade 2 neuropathy
* Valproic acid treatment within 2 weeks of study enrollment
* Systemic steroids, for any indication, stabilized at >10 mg/day prednisone
* Known allergy or hypersensitivity to any component of belinostat, paclitaxel or carboplatin
* Co-existing active infection or any other uncontrolled medical condition likely to interfere with trial procedures
* Active concurrent malignancy (except basal cell carcinoma or cervical intraepithelial neoplasia, other potentially cured malignancy that has been in remission for five years or prior adjuvant therapy for early stage lung cancer that is completed ≥ 12 months ago)
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose ( MTD) of belinostat in combination with carboplatin and paclitaxel in patient with Stage IV non-small cell lung cancer who has received no prior systemic chemotherapy. | 24 Months
  At study entry each eligible patient will be assigned a specific dose level and dose of IV belinostat in mg/m2, to be administered daily on Days 1 to 5 each 21 day cycle, for up to 6 cycles. Dose escalation within each patient is not allowed during this study. At each dose level cohort of up to 6 patients may be evaluated during Cycle 1 of therapy. Multiple dose levels may be evaluated to determine the Maximum Tolerated Dose (MTD) of IV belinostat, in combination with 6 cycles of IV carboplatin and paclitaxel, for chemo-naïve patients with Stage IV NSCLC.

SECONDARY OUTCOMES:
Safety and Tolerability when IV belinostat is administered in combination with carboplatin and paclitaxel in patients with chemotherapy naïve Stage IV M1a or M1b NSCLC. | 24 Months
  Safety will be based on treatment emergent adverse events (TEAEs), including DLTs will be graded by CTCAE version 4.02, and grouped by the MedDRA preferred term, and summarized by worst grade severity per patient. TEAEs are those adverse events that occur or worsen on or after first study treatment up through 30 days post last study treatment, and/or any treatment-related. Tolerability will be mainly characterized by the number and severity of treatment emergent adverse events, and treatment related AEs that occur or worsen after the first dose of study treatment. Deaths, non-fatal serious adverse events (SAEs), and other AEs leading to discontinuation of study treatment will be summarized.
Efficacy when IV belinostat is administered in combination with carboplatin and paclitaxel in patients with chemotherapy naïve Stage IV M1a or M1b NSCLC | 24 Months
  Efficacy variable of this study is best overall response, using RECIST criteria - complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), and not evaluable (NE) - as determined by the investigator.The efficacy endpoint is objective response rate (ORR), defined as the proportion of patients with target lesions who achieve either a CR or a PR.
Progression-free survival (PFS) when IV belinostat is administered in combination with carboplatin and paclitaxel in patients with chemotherapy naïve Stage IV M1a or M1b NSCLC | 24 Months
  progression-free survival (PFS) will be analyzed, defined as the duration of time from date of first study treatment to date of first documented progression or death from any cause. All treated patients will be included in the analysis of PFS. Patients without a documented progression or death will be censored at the last disease assessment.
Objective response rate (ORR) when IV belinostat is administered in combination with carboplatin and paclitaxel in patients with chemotherapy naïve Stage IV M1a or M1b NSCLC. | 24 Months
  The efficacy endpoint is objective response rate (ORR), defined as the proportion of patients with target lesions who achieve either a CR or a PR. A two-sided exact 95% confidence.
  interval (CI) will be calculated for ORR. For example, if 24 patients are to be treated, including 20 patients with target lesions at baseline, and 8 patient achieve a CR or a PR, then the response rate will be 40% with a 95% CI of [19%, 64%].

CONTACTS AND LOCATIONS:
Overall Officials: Brian Matthews, MD, Principal Investigator — Clearview Cancer Institute; Sant Chawla, MD, Principal Investigator — Sarcoma Oncology Center; Saiama Waqar, MD, Principal Investigator — Washington University School of Medicine; Thomas Neiderman, MD, Principal Investigator — University Cancer Insitute
Locations (4):
- United States (4):
  - Clearview Cancer Institute (CCI), Huntsville, Alabama
  - Sarcoma Oncology Center, Santa Monica, California
  - University Cancer Insitute, Boynton Beach, Florida
  - Washington University School of Medicine, St Louis, Missouri